CLINICAL TRIAL: NCT01490515
Title: Embryo Selection Using Non-invasive Metabolomic Analysis Indicates Improvement in Implantation Rates With Fetal Cardiac Activity
Brief Title: Embryo Selection Using Non-invasive Metabolomic Analysis Versus Morphology
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eugonia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: metabolomics
Record Dates: First submitted 2011-12-09; First posted 2011-12-13 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2011-12

CONDITIONS: Embryo Viability
Keywords: non-invasive,; metabolomics,; morphology,; embryo selection,; implantation rates

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Morphology embryo evaluation (Active Comparator): To compare non-invasive metabolomic profiling and the traditional method of morphology assessment for embryo selection in terms of implantation and pregnancy rates in a clinical IVF program.
  Interventions: Other: morphological evaluation
- non-invasive metabolomic profiling (Experimental): To compare non-invasive metabolomic profiling and the traditional method of morphology assessment for embryo selection in terms of implantation and pregnancy rates in a clinical IVF program.
  Interventions: Procedure: non-invasive metabolomic profiling

INTERVENTIONS:
Procedure: non-invasive metabolomic profiling — non-invasive metabolomic profiling of IVF human embryos
  Other Names: ViaMetrics-E, Molecular Biometrics
  Arms: non-invasive metabolomic profiling
Other: morphological evaluation — Simple microscopic observation of embryos and evaluation of morphological characteristics
  Arms: Morphology embryo evaluation

SUMMARY:
Metabolomics was recently introduced in human IVF for non-invasive identification of viable embryos with the highest developmental competence. The investigators intended to investigate if embryo assessment using non-invasive metabolomic profiling leads to increased implantation rates compared to routine morphology evaluation alone.

DETAILED DESCRIPTION:
Metabolomics was recently introduced in human IVF for non-invasive identification of viable embryos with the highest developmental competence. The aim of the present study was to determine whether embryo selection using non-invasive metabolomic profiling as an adjunct to morphology leads to increased implantation rates compared to routine morphology evaluation alone.

ELIGIBILITY:
Inclusion Criteria:

* patients with at least 4 fertilized oocytes

Exclusion Criteria:

* patients with less that 4 fertilized oocytes

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 125 (Actual)
Dates: Start 2010-04; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Implantation rates | 6 weeks of pregnancy
  To compare non-invasive metabolomic profiling and the traditional method of morphology assessment for embryo selection in terms of implantation and pregnancy rates in a clinical IVF program.

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis Sfontouris, PhD, Principal Investigator — Eugonia
Locations (1):
- Eugonia ART Unit, Athens, Attica, Greece

REFERENCES:
- [Background] Scott R, Seli E, Miller K, Sakkas D, Scott K, Burns DH. Noninvasive metabolomic profiling of human embryo culture media using Raman spectroscopy predicts embryonic reproductive potential: a prospective blinded pilot study. Fertil Steril. 2008 Jul;90(1):77-83. doi: 10.1016/j.fertnstert.2007.11.058. Epub 2008 Feb 20. PMID 18281045
- [Background] Seli E, Botros L, Sakkas D, Burns DH. Noninvasive metabolomic profiling of embryo culture media using proton nuclear magnetic resonance correlates with reproductive potential of embryos in women undergoing in vitro fertilization. Fertil Steril. 2008 Dec;90(6):2183-9. doi: 10.1016/j.fertnstert.2008.07.1739. Epub 2008 Oct 8. PMID 18842260
- [Background] Seli E, Sakkas D, Scott R, Kwok SC, Rosendahl SM, Burns DH. Noninvasive metabolomic profiling of embryo culture media using Raman and near-infrared spectroscopy correlates with reproductive potential of embryos in women undergoing in vitro fertilization. Fertil Steril. 2007 Nov;88(5):1350-7. doi: 10.1016/j.fertnstert.2007.07.1390. Epub 2007 Oct 17. PMID 17923129
- [Background] Seli E, Vergouw CG, Morita H, Botros L, Roos P, Lambalk CB, Yamashita N, Kato O, Sakkas D. Noninvasive metabolomic profiling as an adjunct to morphology for noninvasive embryo assessment in women undergoing single embryo transfer. Fertil Steril. 2010 Jul;94(2):535-42. doi: 10.1016/j.fertnstert.2009.03.078. Epub 2009 Jul 8. PMID 19589524
- [Derived] Sfontouris IA, Lainas GT, Sakkas D, Zorzovilis IZ, Petsas GK, Lainas TG. Non-invasive metabolomic analysis using a commercial NIR instrument for embryo selection. J Hum Reprod Sci. 2013 Apr;6(2):133-9. doi: 10.4103/0974-1208.117174. PMID 24082655